CLINICAL TRIAL: NCT03005678
Title: Denosumab Versus Oral Bisphosphonate (Alendronate) for Osteoporosis in Long-term Glucocorticoid Users: an Open Randomized Controlled Trial
Brief Title: Denosumab Versus Bisphosphonates (Alendronate) in GIOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chi Chiu Mok, Principal investigator, Tuen Mun Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC/16
Record Dates: First submitted 2016-12-24; First posted 2016-12-29 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Osteoporosis
Keywords: glucocorticoids, steroids, osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab (Active Comparator): denosumab subcutaneous 60mg every 6 months
  Interventions: Drug: Denosumab
- Alendronate (Placebo Comparator): alendronate 70mg orally every week
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: Denosumab — active treatment group
  Other Names: prolia
  Arms: Denosumab
Drug: Alendronate — comparator
  Other Names: fosamax
  Arms: Alendronate

SUMMARY:
A randomized controlled trial to compare for the efficacy and tolerability of denosumab and oral alendronate in the management of glucocorticoid induced osteoporosis

DETAILED DESCRIPTION:
Study design: an open-label randomized controlled trial Duration of study: 12 months

Treatment arms:

1. Denosumab: a total of 2 doses in a period of 12 months
2. Oral alendronate: weekly dose in a period of 12 months Target sample size: 220 patients (110 patients in each arm)

ELIGIBILITY:
Inclusion Criteria:

1. Adults (women or men) >18 years of age
2. Receiving long-term prednisolone treatment for various medical illnesses, defined as a daily prednisolone dose of ≥2.5mg/day for ≥12 months).
3. Informed consent from patients.
4. Willing to comply with all study procedures

Exclusion Criteria:

1. Patients with previous use of denosumab, teriparatide, intravenous bisphosphonates, strontium or other experimental anti-osteoporotic agents.
2. Premenopausal women who plan for pregnancy within 18 months of study entry.
3. Patients with known bone disorders such as osteomalacia, renal osteodystrophy, and hyperparathyroidism.
4. Patients with unexplained hypocalcemia.
5. Patients with serum creatinine level of >=200umol/L.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
bone mineral density at lumbar spine | month 12
  BMD lumbar spine

SECONDARY OUTCOMES:
bone mineral density at the hip | month 12
  BMD hip
bone turnover markers | month 12
  P1NP and osteocalcin
adverse events | month 12
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: CC Mok, Principal Investigator — Principal Investigator
Locations (1):
- Department of Medicine, Tuen Mun Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No